CLINICAL TRIAL: NCT05610878
Title: Supplementation of Autologous Fat Grafts with Curcumin Preconditioned Adipose-Derived Stem Cells in the Treatment of Facial Contour Deformities
Brief Title: Efficacy of Preconditioned Adipose-Derived Stem Cells in Fat Grafting
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of the Punjab (Other)
Collaborators: Centre of Excellence in Molecular Biology, University of the Punjab, Lahore (Unknown); Higher Education Commission (Pakistan) (Other); Jinnah Burn and Reconstructive Surgery Centre, Lahore (Other Government)
Responsible Party: Principal Investigator, Azra Mehmood, Associate Professor, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEMB-SC01
Record Dates: First submitted 2022-10-26; First posted 2022-11-09 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Romberg Disease; Craniofacial Microsomia; Burn Scar; Post-Traumatic Scar (Disorder)
Keywords: Facial deformities; Fat grafting; Adipose derived stem cells; Preconditioning
MeSH Terms: conditions — Facial Hemiatrophy; Goldenhar Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cultured ASCs enrichment fat grafting (Experimental): Fat graft will be supplemented with naïve ASCs
  Interventions: Biological: Cultured ASCs enrichment fat grafting
- Curcumin-preconditioned ASCs enrichment fat grafting (Experimental): Fat graft will be augmented with curcumin preconditioned ASCs
  Interventions: Biological: Curcumin-preconditioned ASCs enrichment fat grafting
- conventional fat grafting (Active Comparator): Fat graft will not be supplemented with ex-vivo expanded ASCs
  Interventions: Other: Conventional fat grafting

INTERVENTIONS:
Biological: Cultured ASCs enrichment fat grafting — Patients will undergo conventional fat harvesting. Harvested fat will be mixed with cultured ASCs and grafted into recipient site with 1,00,000 cells/ml injected fat
  Arms: Cultured ASCs enrichment fat grafting
Biological: Curcumin-preconditioned ASCs enrichment fat grafting — Patients will undergo conventional fat harvesting. Harvested fat will be mixed with cultured ASCs preconditioned with curcumin and grafted into recipient site with 1,00,000 cells/ml injected fat
  Arms: Curcumin-preconditioned ASCs enrichment fat grafting
Other: Conventional fat grafting — Patients will undergo conventional fat harvesting and grafting of fat into recipient site
  Arms: conventional fat grafting

SUMMARY:
The aim of this study is to evaluate the comparison of therapeutic potential of curcumin preconditioned adipose derived stem cells (ASCs) enrichment fat grafting, naïve ASCs enrichment fat grafting and conventional fat grafting to correct facial contour deformities that cause aesthetic complications in patients.

DETAILED DESCRIPTION:
Human subcutaneous adipose tissue along informed consents will be collected in a lipoaspirate container or 20 cc B.D syringes under the sterilized conditions during the surgery. Fat aspirate collection will be based on certain selection criteria including pre-requisitioning non-diabetic, negative viral status patients. Adipose derived stem cells (ASCs) will be isolated from adipose tissue under sterile aseptic conditions. Firstly, the lipoaspirate container will be opened in the biosafety cabinet and drain off the blood carefully with the help of serological pipette. Then, fat will be washed thrice with 1X phosphate buffer saline (PBS) containing antibiotic and anti-mycotic solution, in order to get rid of blood vessels, hair and other type of connective tissue. After that, the tissue will be enzymatically digested with collagenase type I solution (1mg/ml prepared in Low Glucose Dulbecco's Modified Eagle Medium (LG-DMEM) and incubate for 45 minutes at 37°C on a shaker. After digestion, the enzyme will be inactivated by LG-DMEM augmented with 5% freshly isolated human serum and spin at 1200 rpm for 10 minutes. After centrifugation, fat will be discarded and the infranatant will be passed through 100 µm cell strainers to remove the debris. The filtrate will be centrifuged again for 1200rpm for 8 minutes. Pellet will be resuspended and plated in a sterile T-75 cm2 flask containing 10 ml LG-DMEM supplemented with 5% human serum. The flask will be placed in a humidified incubator at 37°C, 5% carbon dioxide (CO2). The media will be replenished after every third day until the cells got 80-90 % confluency. Cells of P2-P3 stage will be used in this study for immunocytochemistry, and intervention as well. For preconditioning, ASCs will be incubated with curcumin preconditioned medium for 24 h. Cell sterility and viability will be assessed prior to transplantation. For transplantation, 1,00,000 cells per ml of fat will be mixed, transferred to 10 cc syringes and injected at deformity site. Amount of fat will be predetermined by the clinician on the basis of facial asymmetry.

ELIGIBILITY:
Inclusion criteria

* Age 18-50 years (male or female)
* Body-mass index 20-30 kg/m²
* Suitable for liposuction as assessed by the expected cosmetic results
* Provided signed informed consent

Exclusion criteria

* Systemic disorders include autoimmune diseases, hemorrhagic diseases, bone marrow aplasia, sepsis, cancer, and others
* Local disorders include acne, infections and others
* Risk factors include smoking, uncompensated diabetes, hypertension, and allergy to the drugs used for general anesthesia
* Microbiological contamination of either the cell culture or the transplanted tissue

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Volumetric change in facial tissue by ultrasonography | 9 months
  Volumetric evaluation of treated area will be done by measuring the thickness of subcutaneous tissue (in millimeters) by using baseline B mode ultrasound device. Volumetric evaluation of treated area will be done by measuring the thickness of subcutaneous tissue (in millimeters) before transplantation, 1 week after transplantation then after 3, 6 and 9 months by using baseline B mode ultrasound device.

SECONDARY OUTCOMES:
Patient Assessment | 9 months
  Patients will be interviewed and pre-and post-operatively and digital images will be taken until 9 months of follow up.
Surgeon Assessment | 9 months
  Patients will be visually inspected for facial volume by two qualified plastic surgeons unaware of treatment after grafting to check whether curcumin pretreatment have effect on MSCs origin of ASCs.

CONTACTS AND LOCATIONS:
Overall Officials: Azra Mehmood, PhD, Principal Investigator — Center of Excellence in Molecular Biology (CEMB), University of the Punjab, Lahore; Sheikh Riazuddin, PhD, Study Director — Jinnah Burn and Reconstructive Surgery Center (JB&RSC), Lahore
Locations (1):
- Stem Cell Laboratory, Jinnah Burn and Reconstructive Surgery Center (JB&RSC), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Matsumoto D, Sato K, Gonda K, Takaki Y, Shigeura T, Sato T, Aiba-Kojima E, Iizuka F, Inoue K, Suga H, Yoshimura K. Cell-assisted lipotransfer: supportive use of human adipose-derived cells for soft tissue augmentation with lipoinjection. Tissue Eng. 2006 Dec;12(12):3375-82. doi: 10.1089/ten.2006.12.3375. PMID 17518674
- [Background] Bashir MM, Sohail M, Ahmad FJ, Choudhery MS. Preenrichment with Adipose Tissue-Derived Stem Cells Improves Fat Graft Retention in Patients with Contour Deformities of the Face. Stem Cells Int. 2019 Nov 20;2019:5146594. doi: 10.1155/2019/5146594. eCollection 2019. PMID 31827528
- [Background] Ghufran H, Mehmood A, Azam M, Butt H, Ramzan A, Yousaf MA, Ejaz A, Tarar MN, Riazuddin S. Curcumin preconditioned human adipose derived stem cells co-transplanted with platelet rich plasma improve wound healing in diabetic rats. Life Sci. 2020 Sep 15;257:118091. doi: 10.1016/j.lfs.2020.118091. Epub 2020 Jul 12. PMID 32668325
- [Background] Bourne DA, Egro FM, Bliley J, James I, Haas GL, Meyer EM, Donnenberg V, Donnenberg AD, Branstetter B, Coleman S, Rubin JP. Stem Cell Therapy Enriched Fat Grafting for the Reconstruction of Craniofacial Deficits. Plast Reconstr Surg Glob Open. 2023 Jun 19;11(6):e5056. doi: 10.1097/GOX.0000000000005056. eCollection 2023 Jun. PMID 37342306
- [Background] Cao Z, Li H, Wang ZH, Liang XQ. High-Density Fat Grafting Assisted Stromal Vascular Fraction Gel in Facial Deformities. J Craniofac Surg. 2022 Jan-Feb 01;33(1):108-111. doi: 10.1097/SCS.0000000000008038. PMID 34519702
- [Background] Wang C, Long X, Si L, Chen B, Zhang Y, Sun T, Zhang X, Zhao RC, Wang X. A pilot study on ex vivo expanded autologous adipose-derived stem cells of improving fat retention in localized scleroderma patients. Stem Cells Transl Med. 2021 Aug;10(8):1148-1156. doi: 10.1002/sctm.20-0419. Epub 2021 Apr 19. PMID 33871949